CLINICAL TRIAL: NCT05069727
Title: Evaluation of Two Levels of Health Care Interactions in Adolescents With Type 1 Diabetes on Advanced Hybrid Closed Loop System MiniMed 780G/ Zeus Sensor
Brief Title: Simple Initiation of Advanced Hybrid Closed Loop System
Acronym: 780GGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidra Medicine (Other)
Responsible Party: Principal Investigator, Goran Petrovski, Prof MD PhD, Sidra Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 600121
Record Dates: First submitted 2021-09-26; First posted 2021-10-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Diabetes type1
Keywords: Automated Insulin Delivery; Time in Range; Intervention

STUDY DESIGN:
Intervention Model Description: This study is Randomized Clinical Trial, two arm, single-center, clinical investigation in subjects with type 1 diabetes on AHCL insulin pump in a period of 3 months.
  Participants will be randomized in two groups:
  * Group 1, Regular Clinical Protocol, 17 participants
  * Group 2, Simplified Clinical Protocol, 17 participants
Who Masked: Care Provider
Masking Description: Eligible subjects shall be randomly assigned to Group 1 or Group 2 in a 1:1 ratio using a computer-generated randomization scheme developed by the data manager.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, Regular Protocol (Active Comparator): Participants will bolus (insulin), based on carbohydrate content in each meal
  Interventions: Procedure: Regular Protocol with advanced carbohydrate counting
- Group 2, Simplified protocol (Experimental): Participants will bolus (insulin), based on three sets of meal set of meals announcement
  Interventions: Procedure: Simplified Protocol with fixed carbohydrate content

INTERVENTIONS:
Procedure: Regular Protocol with advanced carbohydrate counting — * Review 3 Days CGM data in Manual Mode
  * Carb Ratio by formula 360 / TDD
  * Finetune ICR
  * Target 100 or 110 mg/dl
  * AIT: 2-3 hour
  * Insulin Bolus for meal (advanced carb counting)
  * The parameters will be set using clinical assessment and fine-tuned if needed on F-up visits.
  * Follow up visits will be scheduled Day 7, 14,28, 56 and 84 after enabling SmartGuard (AHCL use).
  Arms: Group 1, Regular Protocol
Procedure: Simplified Protocol with fixed carbohydrate content — * Review 3 Days CGM data in Manual Mode
  * Carb Ratio by formula 360 / TDD ICR 8-10 (TDD 40-60) ICR 5-7 (TDD >60)
  * Target 100 mg/dl
  * AIT: 2 hours
  * Insulin Bolus for meal (Thee sets of meal set of meals announcement carbs will be provided) Regular meal: Total Carbs per Day x 0.6 / 3 Large meal: Total Carbs per Day x 0.6 / 3 x 1.5 Small (Snack) meal: Total Carbs per Day x 0.6 / 3 x 1.5
  * Total carbs per day will be calculated as average on 7-days Food Logbook diary, provided by participant, one week before AHCL initiation.
  * The parameters will be fixed and fine-tuned only in case of hypoglycemia on F-up visits.
  Arms: Group 2, Simplified protocol

SUMMARY:
Background and Aim. The new and advanced hybrid closed loop (AHCL) system MiniMed 780G automatically adjusts basal insulin delivery in addition to automated bolus corrections, based on continuous glucose monitoring (CGM) readings, to offer protection against both hyperglycemia and hypoglycemia.

The objective of this study is to evaluate whether a simplified approach for patients' follow up using preset of pump settings and a simplified meal announcement, followed by minimal interaction can achieve similar glycemic control of AHCL system MiniMed 780G with Guardian Sensor 4 than a regular protocol that is currently used in adolescents with Type 1 Diabetes (T1D).

Methods. This study is Randomized Clinical Trial, two arm, single-center, clinical investigation in subjects with type 1 diabetes on AHCL insulin pump in a period of 3 months. A total of 34 individuals (age 12-18 years) will be enrolled to reach 30 individuals who will complete the 3 months study. Participants will be randomized in two groups: Group 1, Regular Clinical Protocol, 17 participants and Group 2, Simplified Clinical Protocol, 17 participants.

All patients will be recruited during the regular clinic visits to the outpatient Endocrine Clinics at Sidra Medicine in Doha. Patients will be chosen on a first-come first-served basis. Inclusion criteria: Clinical diagnosis of type 1 diabetes, , Age 12-18 years, Basal Bolus therapy >8.0 units per day. Exclusion criteria: Diabetic Ketoacidosis (DKA) in the 6 months prior to screening visit. The initiation protocol consists of four stages: HCL system compatibility assessment, HCL system training, Manual Mode Start and Auto Mode start. Patients will have 7 visits in a period of 3 months after initiation of insulin pump therapy.

Pump initiation: Group 1, Finetune ICR, Target 100 or 110 mg/dl and AIT: 2-3 hour and Group 2, Carb Ratio by formula 360 / TDD, ICR 8-10 (TDD 40-60), ICR 5-7 (TDD >60), Target 100 mg/dl, AIT: 2 hours with fixed meals Results. No group difference in Time in Range (TIR) (70-180mg/dl) > 70% and HbA1c < 7.5% in a period of 3 months after initiation of AHCL.

Conclusion. Conclusions will be drawn on completion of the study and evaluation of the results.

DETAILED DESCRIPTION:
This study is Randomized Clinical Trial, two arm, single-center, clinical investigation in subjects with type 1 diabetes on AHCL insulin pump in a period of 3 months.

A total of 34 individuals (age 12-18 years) will be enrolled to reach 30 individuals who will complete the 3 months study.

Participants will be randomized in two groups:

* Group 1, Regular Clinical Protocol, 17 participants
* Group 2, Simplified Clinical Protocol, 17 participants Intervention Description
* Intervention in Group 2, Simplified protocol.
* Insulin Carb Ratio (ICR) by formula 360 / Total Daily Dose (TDD)

  * ICR 8-10 (TDD 40-60)
  * ICR 5-7 (TDD >60)
* Target 100 mg/dl
* Active Insulin Time (AIT): 2 hours
* Meals: Thee sets of meal set of meals announcement carbs calculated by the following formula:

  * Regular meal: Total Carbs per Day x 0.6 / 3
  * Large meal: Total Carbs per Day x 0.6 / 3 x 1.5
  * Small (Snack) meal: Total Carbs per Day x 0.6 / 3 x 1.5 * Efficacy The efficacy shall be measured Time in Ranges (provided by CGM data), for Time in Range (70-180mg/dl), Time below Range(<70mg/dl) and Time above Range (>180 mg/dl) in the third month of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes >0.5 year prior to consent date. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. Age 12-18 years and above at the initiation of the system
3. Total daily insulin use of great than 8.0 units per day over a 1-week period
4. Willing and able (access to internet from home)
5. Clinically able to start the AHCL system

Exclusion Criteria:

1. Pregnancy
2. Untreated diabetes retinopathy, or other causes that in the investigator's opinion , precludes the individual from participating in the trial.
3. Currently in other Clinical Trial

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Time in Range( 70-180 mg/dl) | Third month
  Group change in the third month of AHCL use

SECONDARY OUTCOMES:
HbA1c | 3 months
  Change between groups
Average Sensor Glucose | 3 months
  Change between groups
Time Bellow Range (<70 mg/dl, <54 mg/dl) | 3 months
  Change between groups
Time Above Range (>180 mg/dl) | 3 months
  Change between groups
Diabetic Ketoacidosis | 3 months
  Number of events in each group
Severe Hypoglycemia | 3 months
  Number of events in each group

OTHER OUTCOMES:
Sensor wear | 3 months
  % of sensor wear, change between each groups
Auto Mode - SmartGuard | 3 months
  % of Automode-SmartGuard, change between groups
Total Daily Insulin | 3 months
  % of Automode, Change between each groups

CONTACTS AND LOCATIONS:
Overall Officials: Goran Petrovski, PhD, Principal Investigator — Sidra Medicine
Locations (1):
- Sidra Medicine, Doha, Qa, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrovski G, Al Khalaf F, Campbell J, Fisher H, Umer F, Hussain K. From Multiple Daily Injections to Hybrid Closed-Loop System in Ten Days, Utilizing a Structured Initiation Protocol. J Diabetes Sci Technol. 2020 May;14(3):689-690. doi: 10.1177/1932296819895509. Epub 2019 Dec 26. No abstract available. PMID 31876178
- [Result] Bergenstal RM, Nimri R, Beck RW, Criego A, Laffel L, Schatz D, Battelino T, Danne T, Weinzimer SA, Sibayan J, Johnson ML, Bailey RJ, Calhoun P, Carlson A, Isganaitis E, Bello R, Albanese-O'Neill A, Dovc K, Biester T, Weyman K, Hood K, Phillip M; FLAIR Study Group. A comparison of two hybrid closed-loop systems in adolescents and young adults with type 1 diabetes (FLAIR): a multicentre, randomised, crossover trial. Lancet. 2021 Jan 16;397(10270):208-219. doi: 10.1016/S0140-6736(20)32514-9. PMID 33453783
- [Result] Beato-Vibora PI, Gallego-Gamero F, Ambrojo-Lopez A, Gil-Poch E, Martin-Romo I, Arroyo-Diez FJ. Rapid Improvement in Time in Range After the Implementation of an Advanced Hybrid Closed-Loop System in Adolescents and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2021 Sep;23(9):609-615. doi: 10.1089/dia.2021.0037. Epub 2021 Apr 20. PMID 33784187
- [Result] Lee MH, Vogrin S, Paldus B, Jones HM, Obeyesekere V, Sims C, Wyatt SA, Ward GM, McAuley SA, MacIsaac RJ, Krishnamurthy B, Sundararajan V, Jenkins AJ, O'Neal DN. Glucose Control in Adults with Type 1 Diabetes Using a Medtronic Prototype Enhanced-Hybrid Closed-Loop System: A Feasibility Study. Diabetes Technol Ther. 2019 Sep;21(9):499-506. doi: 10.1089/dia.2019.0120. Epub 2019 Jul 2. PMID 31264889
- [Result] Paldus B, Lee MH, Jones HM, McAuley SA, Horsburgh JC, Roem KL, Ward GM, MacIsaac RJ, Cohen N, Colman PG, Jenkins AJ, O'Neal DN. Glucose Control Using a Standard Versus an Enhanced Hybrid Closed Loop System: A Randomized Crossover Study. Diabetes Technol Ther. 2019 Jan;21(1):56-58. doi: 10.1089/dia.2018.0279. PMID 30620641
- [Result] Petrovski G, Al Khalaf F, Campbell J, Fisher H, Umer F, Hussain K. 10-Day structured initiation protocol from multiple daily injection to hybrid closed-loop system in children and adolescents with type 1 diabetes. Acta Diabetol. 2020 Jun;57(6):681-687. doi: 10.1007/s00592-019-01472-w. Epub 2020 Jan 17. PMID 31953687
- [Derived] Petrovski G, Campbell J, Pasha M, Hussain K, Khalifa A, Umer F, Almajaly D, Hamdar M, Heuvel TVD, Edd SN. Twelve-Month Follow-up from a Randomized Controlled Trial of Simplified Meal Announcement Versus Precise Carbohydrate Counting in Adolescents with Type 1 Diabetes Using the MiniMed 780G Advanced Hybrid Closed-Loop System. Diabetes Technol Ther. 2024 Mar;26(S3):76-83. doi: 10.1089/dia.2023.0429. PMID 38377327